CLINICAL TRIAL: NCT03333889
Title: Patient Satisfaction and Crestal Bone Loss of Polymer Infiltrated Ceramic Network Versus Lithium Disilicate Implant Hybrid Abutment Crowns in Esthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Inas Adel Mahmoud, assistant lecturer,fixed prosthodontic department, faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-11-02
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Hybrid Crowns on Single Implants in Esthetic Zone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind :outcome asessor,participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-max hybrid crown (Active Comparator): E-max hybrid crown Lithium Disilicate based ceramic which is characterized by high strength and optimum esthetics and considered a gold standard in anterior restorations
  Interventions: Other: emax hybrid crown
- Vita Enamic hybrid crown (Experimental): Vita Enamic hybrid crown polymer infilltrated ceramic network(hybrid ceramic) characterized by low modulus of elasticity that acts as cushion on implants.
  Interventions: Other: Vita Enamic hybrid crown

INTERVENTIONS:
Other: Vita Enamic hybrid crown — hybrid ceramic material in the form of mesoblocks where the ceramic block is attached to a ti base .The whole assembly is screw retained superstructure.
  Arms: Vita Enamic hybrid crown
Other: emax hybrid crown — high srength glass ceramic that can be milled in sections up to 1mm .
  Arms: E-max hybrid crown

SUMMARY:
P: Population: Patients requiring single unit implant restoration in esthetic zone I: Intervention: Polymer-infiltrated-ceramic-network abutment crown (VITA Enamic-VITA Zahnfabrik) C: Comparison: Lithium disilicate ceramic abutment crown (IPS e. max-Ivoclar Vivadent) O: Outcome: patient satisfaction , crestal bone loss and periodontal parameters T: Time: 12 months S :Randomized controlled trial research question:For patients receiving implants in esthetic zone, Does the use of polymer-infiltrated-ceramic-network hybrid abutment crown offer better patient satisfaction , less bone loss and better peri-implant clinical parameters when compared to lithium disilicate hybrid abutment crowns?

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years old.
2. Patients able to read and sign the informed consent document.
3. Medically free patients or with controlled systemic disease.
4. Patients with good bone quality and quantity evaluated using C.B.C.T.
5. Patients willing to return for follow-up examinations and evaluation.
6. Patients having single missing recently extracted premolar tooth.

Exclusion Criteria:

1. Young patients in growth stage.
2. Patients with unsuitable implantation sites (patients with major boney defects or sever bone resorption)
3. Pregnant women to avoid any complication that may occur in dental office.
4. Patients with uncontrolled systemic disease (hypertensive patient or uncontrolled diabetic patient)
5. Psychiatric problems or unrealistic expectations.
6. Multiple adjacent missing teeth.
7. Patients with bad oral hygiene. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 12 months
  using visual analogue scale (o-unsatisfied up to max 10 satisfied)

SECONDARY OUTCOMES:
crestal bone loss | 12 months
  using digital subtraction technique

CONTACTS AND LOCATIONS:
Locations (1):
- Inas adel mahmoud, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided